CLINICAL TRIAL: NCT04350749
Title: Platelet Rich Fibrin (PRF) Membranes in Lateral Alveolar Ridge Augmentation. A Randomized Controlled Study Comparing an Autogenous Bone Graft Covered by a Platelet Rich Fibrin (PRF) Membrane (Test Group) or an Anorganic Bovine Bone Substitute and a Resorbable Collagen Barrier Membrane (Control Group)
Brief Title: The Use of Platelet-rich Fibrin (PRF) Membranes in Lateral Alveolar Ridge Augmentation When Jaw Bone is Missing Before Dental Implant Installation. A Study Comparing an Autogenous Bone Block Graft Covered Either by a (PRF) Membrane (Test) or Bone Substitute and a Barrier Membrane (Control)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Boneaugmentation1234
Record Dates: First submitted 2020-04-05; First posted 2020-04-17 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Tooth-loss
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: Clinical randomized controlled trial
Masking Description: Some of the data anlysis is masked. The examiner is blinded when performing the CBCT scan analysis of the volume (Study 2) and the histological assessment of the bone biopsies (Study 3)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (PRF group) (Experimental): PRF membrane is added to the bone block to evaluate if any effect on bone healing, soft healing, post-operativ pain
  Interventions: Biological: PRF is added in the test group.
- Control group (Standard operation) (Active Comparator): A standard bone augmentation procedure, which is weel-described is performed to compare the outcome of the test group
  Interventions: Biological: PRF is added in the test group.

INTERVENTIONS:
Biological: PRF is added in the test group. — The PRF membrane can be considered as a biological membrane

SUMMARY:
Tooth loss can in many cases be treated with an artificial titanium root (dental implant) and subsequent manufacture of a porcelain crown. After the tooth is lost bone resorption of the existing jaw bone often occurs making implant placement difficult. Therefore, bone augmentation is often necessary before implant placement. Six months after the bone augmentation has been performed, the implant can be inserted into the jaw bone and after additionally 6 months the final porcelain crown can be mounted.

Reconstruction of the jaw bone is often done by harvesting a bone block from the patient's own jaw. The bone block is harvested typically from the posterior part of the lower jaw, where after it is placed and fixated by screws in the part of the jaw where the bone is missing. Finally, the bone graft is covered with artificial bone substitute and a collagen membrane. Recent studies have suggested that adding platelet-rich fibrin (PRF) membranes will have an advantageously effect in reconstruction of the jaw bone and bone healing. PRF membranes are derived from a blood sample of the patient and has been introduced to accelerate soft tissue as well as bone healing. No comparative studies have been conducted in humans for the time being evaluating the effect of PRF in conjunction with bone augmentation. Therefore, the purpose of this study is to compare a control group with a test group in which the control group is treated in a standardized manner, while PRF is added to the bone graft in the test group. After 6 months of bone healing, a dental implant can be inserted in both groups using a standard technique.

For the two groups, the following is examined:

1. The final treatment outcome of the dental implant focusing on clinical outcome, radiologic outcome, aesthetic outcome, patient satisfaction.
2. Bone changes over time with a focus on volume changes. In addition, focus on soft tissue healing.
3. Bone healing assessed using bone biopsies taken in connection with the implant installation.

All included patients is missing a tooth where bone augmentation is needed before an implant can be inserted. A general study is conducted and patients are randomly assigned to a control group (20 patients) and a test group (20 patients). The control group is treated with a standard bone augmentation procedure. This is done in local anesthesia, where initially a bone graft is removed from the back of the lower jaw. The gingiva corresponding to the toothless area is loosened and the bone graft is fixed with 2 titanium screws before being covered with a artificial bone substitute and a membrane to protect the bone graft during the healing period. The test group is treated in the same way, however, a PRF-membrane is used instead of the bone substitute material and the membrane. The PRF-membrane is prepared by taking a blood sample from the arm (80 ml) as with a regular blood sample. The blood is centrifuged, which transforms the blood into a platelet-rich membrane. Thus, the membrane is produced 100% natural without any additives. However, the membranes contain growth factors that have the potential to promote mucosal and bone healing. In both groups, common penicillin (Amoxicillin / Clavulanic acid, 1000/250 mg) and painkillers (Ibuprofen, 400 mg x 4, supplemented with Panodil 1000 mg x 4) are given before surgery.

After six months, the dental implant is inserted using standard procedure in both groups. The gingiva is set aside and perpendicular to the bone grafted area, a cylindrical bone tissue biopsy (2 mm in diameter, approximately 8 mm long) is taken containing the applied bone graft and the original jaw comb (for study 3). Then the previously inserted 2 titanium screws are removed and the implant is inserted.

After another six months, the final porcelain crown is made. The implant is exposed and a healing cap is applied. After 2-3 weeks, the gum is healed, after which the final impression is made to the crown, which the patient will have installed 1-2 weeks after.

The bone augmentation procedure, the implant installation and manufacturing of the porcelain crown are characterized by minimal risks and complications. In bone augmentation, there is minimal risk of altered sensation similar to the lower lip. It is typically of a temporary nature but can be permanent in very rare cases. The implant operation, including subsequent crown manufacturing, is performed in both groups by a standardized procedure, which is also characterized by minimal risk of side effects and complications. Thus, numerous studies have shown that implant treatment is characterized by a high implant survival of approx. 95% after 10 years.

As part of the treatment, a total of 3 scans of the jaw (for study2) as well as 3 ordinary dental films are made for assessment of the jaw bone volume and as a control of the bone around the implant. This radiation dose equals approximately 60 days of background radiation in Denmark.

DETAILED DESCRIPTION:
Project title: Platelet rich fibrin (PRF) membranes in lateral alveolar ridge augmentation.

Background Tooth loss induce extensive resorption of the alveolar ridge, thereby compromising implant placement in a correct anatomical position. Therefore, various procedures for alveolar ridge augmentation have been introduced. The most frequently used procedure includes lateral alveolar ridge augmentation by an autogenous bone graft harvested from an intraoral donor site. The bone graft is often covered by a resorbable collagen barrier membrane and an anorganic bovine bone substitute to minimize the resorption of the autogenous bone graft during the healing period. However, it has been indicated that the use of a barrier membrane increases the risk of bone graft exposure, thereby significantly compromising the treatment outcome.

Biological platelet rich fibrin (PRF) membranes derived from a blood sample of the patient has been introduced to accelerate soft tissue as well as bone healing. In vitro studies have revealed that PRF membranes may enhance proliferation and differentiation of osteoblasts, collagen protein production, and angiogenesis. The potential benefit of PRF membranes for lateral alveolar ridge augmentation has been evaluated in one animal experiment only. However, the use of PRF membranes in lateral alveolar ridge augmentation has not been addressed in humans. Clinical studies using PRF membranes have indicated accelerated soft tissue and bone healing in periodontal therapy, soft tissue reconstructive surgery, and vertical alveolar ridge augmentation using the maxillary sinus lift procedures.

Purpose of investigations, including hypothesis

The purpose of the investigations is to evaluate the treatment outcome after lateral alveolar ridge augmentation by using an autogenous bone graft covered by 1) a PRF membrane (test group) or 2) an anorganic bovine bone substitute and a resorbable collagen barrier membrane (control group) in a randomized, controlled clinical trial (RCT) with focus on:

Study 1: Outcome of the oral implant treatment with focus on clinical, radiographic, esthetic, and socioeconomical parameters.

Study 2: Soft tissue and bone healing with focus on volumetric changes. Study 3: Bone healing by using histological and stereological methods. It is the investigator's hypothesis that there are no differences between the test and control groups.

Material and methods A total of 40 patients with a healthy dentition are included at random within the test (n=20) and control (n=20) group in the study.

Lateral alveolar ridge augmentation The lateral alveolar ridge augmentation is performed as previously described. An autogenous bone graft is initially harvested from the mandible via an intraoral approach. The lateral aspect of the posterior part of the mandible is exposed by using a standard incision technique and the harvested bone graft is adjusted and fixated with two titanium mini-screws as a lateral block graft. In the test group, a venous blood sample (80 ml) via puncture of a vein in the fossa cubiti is collected and centrifuged according to a previously described method. A total of 20 ml of the 80 ml collected blood is collected for later biochemical characterization of the blood sample and the PRF membrane. The obtained PRF membrane is adjusted and placed to cover the bone graft. In the control group, the lateral block graft is covered with anorganic bovine bone substitute (Bio-Oss, Geistlich Pharma, Switzerland) and a collagen membrane (Bio-Gide, Geistlich Pharma, Switzerland). Preoperative prophylactic antibiotic treatment (Amoxicillin/Clavulanic acid, 1000/250 mg) is given as well as postoperative pain control (Ibuprofen, 400 mg x 4 daily).

Implant installation After a healing period of 6 month, a standard incision technique is used to expose the augmented alveolar ridge. The previously inserted mini-screws are removed and an implant (Bone Level, Straumann, Switzerland) with a cover screw is installed according to the manufacture's recommendation. Before implant installation, a cylindrical biopsy of the augmented bone and the resident alveolar bone is retrieved perpendicularly to the lateral aspect of the augmented ridge by a 2-mm trephine bur for later histological and stereological evaluation. The biopsy cavity is filled with locally harvested autogenous bone chips (Safescraper, Divisione Medical Meta, Italy). If the buccal bone thickness after implant installation is less than 2 mm, localized alveolar ridge augmentation is performed by using also locally harvested autogenous bone chips covered by an anorganic bovine bone substitute and a resorbable collagen membrane. Preoperative prophylactic antibiotic treatment (Amoxicillin/Clavulanic acid, 1000/250 mg) is given as well as postoperative pain control (Ibuprofen, 400 mg x 4 daily).

Prosthetic treatment After a healing period of 6 month, a healing abutment is placed (Nobel Biocare, Switzerland). After an additional 2-week soft tissue healing period, the healing abutment is removed and an individual definitive zirconium abutment and an all-ceramic crown with a framework of alumina oxide and veneering porcelain is placed.

Data analysis, including calculation of sample size Data management and analysis including calculation of descriptive statistics are performed in collaboration with a biostatistician. The statistical analyses will mainly include t-test, Pearson's correlation analysis, and analysis of variance. Power calculations are based on differences in patient satisfaction and changes in marginal bone level in a previous study involving replacement of a single tooth with 2 different protocols of implant treatment. When the calculation of the group size is based on the figures for patient satisfaction measured on a VAS scale (with a maximum of 100) after treatment (a difference between treatments of 6.81 and a standard deviation of 6.82), 17 patients should be included in each group to detect a difference at the 5%-level with a power of 80%. When the power calculation is based on the observed changes in marginal bone level from insertion of the implant to abutment connection (a change of 0.65 mm and a standard deviation of 0.65), 17 patients in each group reaches a power of 97% at the 5%-level. With 15% to cover any drop-outs, each treatment group should include 20 patients.

Bone biopsy storage The previously describes bone biopsies are kept during the histological processing at Aarhus University. All material will be anonymous and destroyed at the end of the project.

Ethical aspects, including risks, data management, and publication The two described lateral alveolar ridge augmentation procedures are both commonly used in the clinic. As previously described, potential benefits and disadvantages are presently unknown, because no comparative study has been performed. The described implant treatment is performed according standard procedure. It has been documented that lateral alveolar ridge augmentation and implant treatment are characterized by minimal risk of complication, including pain, swelling, and inflammation. The bone harvesting procedure includes a minimum risk for compromised sensibility of the lip and tongue. The change in sensibility is in most cases temporarily, but can rarely be permanent. The study involves a total of 3 segmented CBCT scanning procedures and 5 intra-oral radiographic images corresponding to a total radiation dose equivalent to 60 days of background radiation. Therefore, the total radiation dose of the patients seems from an ethical point of view acceptable. In conclusion, the described study is characterized by a very low risk of complications. If failure of the augmentation procedure or implant treatment occurs, prosthetic treatment involving a conventional, fixed bridge can always be performed. If unexpected adverse events occur, the project will be cancelled.

The all surgical procedures will be performed by the applicant, who is an oral and maxillofacial surgeon with extensive clinical skills within the field of bone augmentation and implant treatment. Moreover, the prosthetic part of the treatment will be performed by two dentists with extensive clinical skills within the field of implant prosthetics. The patients will be covered by the same health assurance as all patients at the Department of Dentistry, Aarhus University.

PRF membranes derived from the patient's own blood using a chair-side method have recently been commercially available. These membranes may enhance soft tissue as well as bone healing, but the hypothesis has not been validated in a randomized controlled clinical trial. The described studies will provide new and important knowledge, which from a clinical, economical, and scientific perspective is important.

The studies are performed according to the Declaration of Helsinki and internationally accepted guidelines for randomized controlled clinical trials (RCT), and has been approved in accordance with Danish regulations by the Committee of Ethics, the Central Denmark Region (Project-ID: 44710) 2014 before the start of the study. The physical and mental integrity of the patients will be respect. The project is performed as Ph.D. collaboration project between Aarhus University and Aarhus University Hospital after approval by the Danish Data Protection Agency. All processing of personal data and free movement of such data will be in according to Danish law. The results will be published in international scientific journals.

Funding The project has been developed by the applicant in collaboration with the supervisors without commercial influences. Aarhus University has supported the project and used material including implants will be provided for free by the manufactures (Nobel Biocare and Geistlich Pharma, Switzerland). These companies will not have any influence on the project, including publication of the results.

The patients are recruited among patients referred to the Department of Dentistry, Aarhus University from dentist for bone augmentation and implant treatment. If insufficient numbers of patients are referred, advertisement of the project will be announced by e-mail or within the Danish Dental Journal (Tandlægebladet). Detailed written and oral information about the project including all potential risks will be given by the applicant in a separate, undisturbed clinic at the Section for Oral and Maxillofacial Surgery and Oral Pathology, Department of Dentistry, Aarhus University. The patients will be provided with the written information at the time of the initial examination. All patients will have sufficient time to read the information before the oral information is given. Moreover, the patients will be given sufficient time (1 week) to consider their participation in the study before the informed consent form is signed and dated by the patient as well as the applicant. The patients will receive the original version, while the applicant will keep a copy as part of the study documentation. The patients are provided with the opportunity to have an assessor during the entire information and approval phase.

The patients will be treated at the Department of Dentistry, Health, Aarhus University and the Department of Oral and Maxillofacial Surgery, Aarhus University Hospital, Denmark.

ELIGIBILITY:
Inclusion Criteria:

Tooth loss Atrophy of the alveolar process.

Exclusion Criteria:

Oral pathology Bruxism. Allergies to bovine and porcine biomaterials

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Difference of volumetric bone changes of the augmented bone 6 month after the primary bone augmentation procedure between the test and control group | 6 month after the primary bone augmentation procedure
  The change of the augmented bone volume is assessed by comparing CBCT scans at different timepoint: Baseline=Before bone augmentation;After bone augmentation=Immediate after bone augmentation; Follow-up= Prior to implant installation (6 month after the primary bone augmentation). The volumetric bone changes over time were calculated as bone resorption rate, i.e. the difference in bone volume two weeks after bone augmentation and bone volume 6 months after augmentation.
Difference of the various tissue component of the augmented bone between the test and control group | 6 month after the primary bone augmentation procedure (in the same phase as the implant installation).
  A cylindrical biopsy of the augmented region is retrieved perpendicularly to the lateral aspect of the augmented bone 6 month after the primary bone augmentation (in the same surgical phase as the implant installation). The bone biopsies are evaluated by histological and histomorphometric analyses with focus on vital bone, non-vital bone, soft tissue, and blood vessels
Difference of implant survival between the test and the control group | Final follow-up 12 month after the implant supported crown is mounted (24 month after the primary bone augmentation)
  Implant survival is registered at the final follow-up. Implant failure is defined as clinically visible implant mobility or removal of a stable implant due to progressive peri-implant bone loss or infection.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Erik Noerholt, DDS, Principal Investigator — University of Aarhus
Locations (1):
- Department of Dentistry and Oral Health, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartlev J, Schou S, Isidor F, Norholt SE. A clinical and radiographic study of implants placed in autogenous bone grafts covered by either a platelet-rich fibrin membrane or deproteinised bovine bone mineral and a collagen membrane: a pilot randomised controlled clinical trial with a 2-year follow-up. Int J Implant Dent. 2021 Feb 8;7(1):8. doi: 10.1186/s40729-021-00289-z. PMID 33554323